CLINICAL TRIAL: NCT06639984
Title: Assessing Psyllium Given With Meals for Fructan Sensitivity in Children With Irritable Bowel Syndrome
Brief Title: Psyllium in Pediatric IBS
Acronym: Psyllium
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dr Bruno Chumpitazi, M.D. (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Dr Bruno Chumpitazi, M.D., Instructor Temporary in the Department of Pediatrics, Pediatrics, Gastroenterology, Hepatology and Nutrition, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00114630
Record Dates: First submitted 2024-09-25; First posted 2024-10-15 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-03

CONDITIONS: Irritable Bowel Syndrome
Keywords: Abdominal Pain
MeSH Terms: conditions — Irritable Bowel Syndrome; Abdominal Pain | interventions — Psyllium; Fructans

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Psyllium (0.7 g/year of age per day) given with fructans (Active Comparator): Participants will receive Psyllium (0.7 g/year of age per day) given with fructans (daily dose 0.5 g/kg up to 19 grams)
  Interventions: Drug: Psyllium (0.7 g/year of age per day); Other: fructans
- Psyllium (0.5 g/year of age per day) given with fructans (Active Comparator): Participants will receive Psyllium (0.5 g/year of age per day) given with fructans (daily dose 0.5 g/kg up to 19 grams)
  Interventions: Drug: Psyllium (0.5 g/year of age per day); Other: fructans
- Placebo (0.7 g/year of age glucose) given with fructans (Placebo Comparator): Participants will receive Placebo (0.7 g/year of age glucose) given with fructans (daily dose 0.5 g/kg up to 19 grams).
  Interventions: Drug: Placebo; Other: fructans

INTERVENTIONS:
Drug: Psyllium (0.7 g/year of age per day) — Psyllium (0.7 g/year of age per day) (Konsyl Pharmaceuticals, Easton, MD)
  Arms: Psyllium (0.7 g/year of age per day) given with fructans
Drug: Psyllium (0.5 g/year of age per day) — Psyllium (0.5 g/year of age per day) (Konsyl Pharmaceuticals, Easton, MD)
  Arms: Psyllium (0.5 g/year of age per day) given with fructans
Drug: Placebo — Placebo (0.7 g/year of age glucose) (Staleydex 333; Tate & Lyle, Staley, London, UK)
  Arms: Placebo (0.7 g/year of age glucose) given with fructans
Other: fructans — Daily dose 0.5 g/kg up to 19 grams, Orafti Synergy1

SUMMARY:
The goal of this clinical trial is to learn if a fiber (psyllium) can change the way bacteria use fructans (a type of sugar) and whether psyllium can help decrease childhood irritable bowel syndrome (IBS) symptoms when eating fructans. The main questions it aims to answer are:

Aim 1: The effect of psyllium at two doses given with a fructan meal on microbial fructan fermentation (intracolonic pH; H2 gas production; gut microbiome composition; fecal short-chain fatty acids, lactate, glycomics).

Aim 2: Determine the impact of psyllium given with a fructan meal on fructan-induced GI symptoms.

Participants will first be asked to eat a specific diet over two three-day periods to determine if fructans worsen their IBS symptoms. Those with worsening symptoms with fructans will be asked to participate in the second part of the study. This includes two weeks of baseline (no change in diet) and two weeks of eating a specific diet with fructans with either psyllium or glucose. Participants will be asked to complete pain and stool diaries, submit stool specimens, swallow a pill to capture gut acid levels, and give breath samples.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 12-17 years meeting pediatric Rome IV criteria for IBS

Exclusion Criteria:

* Children who have had previous bowel surgery, have documented GI disorders (e.g., ulcerative colitis), or a serious chronic medical condition (e.g., diabetes)
* weight and/or height are > or < 2 SD for age
* have chronic conditions with GI symptoms (e.g., cystic fibrosis)
* have been on antibiotics or probiotics within 3 months (because of potential alterations to the GI microbiome0
* girls who are pregnant (tested with urine beta-human chorionic gonadotropin at the initial visit)

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in microbiome composition measured via taxonomic profiling using 16S ribosomal RNA gene amplicon sequencing | Baseline, 2 weeks
Change in fecal lactate | Baseline, 2 weeks
Change in fecal short-chain fatty acids | Baseline, 2 weeks
Change in hydrogen gas production | Baseline, 2 weeks
Change in fecal fructans | Baseline, 2 weeks

SECONDARY OUTCOMES:
Change in abdominal pain frequency | Baseline, 2 weeks
Change in abdominal pain severity | Baseline, 2 weeks
  Participants will rate abdominal pain on a scale of 0-10, with higher scores indicating more severe pain.
Change in bloating severity | Baseline, 2 weeks
  Participants will rate bloating on a scale of 0-10, with higher scores indicating worse bloating.
Change in flatulence severity | Baseline, 2 weeks
  Participants will rate flatulence on a scale of 0-10, with higher scores indicating worse flatulence.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Chumpitazi, MD, MPH, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No